CLINICAL TRIAL: NCT05313815
Title: Moderate Hypofractionated Boost to the Prostate With Pelvic RT in High Risk Prostate Cancer
Acronym: MOB-RT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5218
Record Dates: First submitted 2022-03-15; First posted 2022-04-06 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; high risk prostate cancer; high-risk prostate cancer; node positive prostate cancer; nod-positive prostate cancer; hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderate Hypofracitonated Boost to the Prostate with Pelvic Radiation Therapy (Experimental): External beam radiotherapy- 60 Gy in 20 fractions to the prostate, 48 Gy in 20 fractions to the pelvis, 68 Gy in 20 fraction optional boost to prostatic dominant intraprostatic lesion, 55 Gy in 20 fraction optional boost to involved pelvic lymph nodes
  Interventions: Radiation: Moderate hypofractionated boost to the prostate with pelvic RT (external beam radiotherapy)

INTERVENTIONS:
Radiation: Moderate hypofractionated boost to the prostate with pelvic RT (external beam radiotherapy) — External beam radiotherapy- 60 Gy in 20 fractions to the prostate, 48 Gy in 20 fractions to the pelvis, 68 Gy in 20 fraction optional boost to prostatic dominant intraprostatic lesion, 55 Gy in 20 fraction optional boost to involved pelvic lymph nodes

SUMMARY:
This is a single-arm phase II prospective trials that is recruiting 100 participants. The study population that is being investigated are patients with localized high-risk or node-positive prostate cancer. Participants will receive external beam radiotherapy as a moderately hypofractionated boost to the prostate with pelvic radiation therapy. Androgen deprivation therapy will be prescribed at the discretion of the treating physician as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Able to provide informed consent.
* Histologic diagnosis of prostate adenocarcinoma.
* ECOG performance status 0-1.
* High-risk localized disease by NCCN criteria (>cT3, Grade group >4, or PSA >20 ng/mL) or clinical N1 disease.
* Clinical M0 by conventional imaging (computed tomography (CT) and bone scan (BS)) and/or molecular imaging (prostate specific membrane antigen (PSMA)- positron emission tomography (PET))

Exclusion Criteria:

* Prior pelvic radiotherapy.
* Contraindications to radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Acute Grade >2 Gastrointestinal Toxicity | Baseline to 5-year follow-up
  Acute (less than or equal to 90 days) toxicity will be evaluated by using prospective follow-up and grading according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Patient-reported quality-of-life assessed by EPIC-26 | Baseline to 5-year Follow-up
  Patient-Reported Quality of Life will be assessed at baseline and at each follow-up visit (3-weeks post intervention then every 6 months until 5 years, or more frequently if clinically necessary) using the following assessment questionnaires: 26-Item Expanded Prostate Cancer Index Composite (EPIC-26)
Measure the severity of lower urinary tract symptoms during the study | Baseline to 5-year Follow-up
  Patient-Reported symptoms will be assessed at baseline and at each follow-up visit (3-weeks post intervention then every 6 months until 5 years, or more frequently if clinically necessary) using the following assessment questionnaires: International Prostate Symptom Score (IPSS)
Graded criteria based on CTCAE version 5.0 for acute genitourinary toxicity and late genitourinary and gastrointestinal toxicity | Baseline to 5-year Follow-up
  Acute (less than or equal to 90 days) and long-term (greater than 90 days) toxicity will be evaluated by using prospective follow-up and grading according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Measure of oncologic outcomes | Baseline to 5-year Follow-up
  Time to development of castrate-resistant prostate cancer (biochemmical or ardiographic progression while having castrate levels of testosterone)
Measure of oncologic outcomes | Baseline to 5-year Follow-up
  Biochemical control rate will be assessed at baseline and at each follow-up visit (3 weeks after treatment then every 6 months until 5 years or more frequently if clinically necessary) by the blood level of prostate-specific antigen (PSA) levels
Measure of onocologic outcomes | Baseline to 5-year Follow-up
  Radiographic control rate will be assess at baseline and weekly during the radiotherapy intervention using cone beam CT or bone scan.
Prostate cancer specific survival based on death from prostate cancer | Baseline to 5-year Follow-up
  Safety will be evaluated by recording prostate cancer mortality at follow-up visits (3-weeks post intervention then every 6 months until 5 years, or more frequently if clinically necessary)
Overall survival | Baseline to 5-year Follow-up
  Safety will be evaluated by recording overall mortality at follow-up visits (3-weeks post intervention then every 6 months until 5 years, or more frequently if clinically necessary).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada